CLINICAL TRIAL: NCT04978961
Title: A Novel Treatment Delivery of Acceptance and Commitment Therapy for Chronic Pain in an Integrated Primary Care Setting
Brief Title: Acceptance and Commitment Therapy for Chronic Pain in Integrated Primary Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HSC20160512H
Record Dates: First submitted 2021-07-15; First posted 2021-07-27 (Actual); Last update posted 2021-07-27 (Actual); Status verified 2021-07

CONDITIONS: Chronic Pain
Keywords: chronic pain; acceptance and commitment therapy; integrated primary care; behavioral health consultant
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Masking Description: PI was masked to assessment outcomes during intervention phase
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Focused Acceptance and Commitment Therapy (FACT) (Experimental): Focused Acceptance & Commitment Therapy (FACT): FACT is a brief type of cognitive behavioral therapy that helps patients reduce disability through increased acceptance, reconnection with values, and reduced unhelpful control/coping strategies. Patients randomized to the intervention group received FACT per the study manual, delivered by an integrated Behavioral Health Consultant (BHC). Patients had one individual visit (30 minutes) and three consecutive weekly group visits (one hour) followed by a booster visit two months later. These classes (group visits) were rolling, not cohort-driven, meaning new and returning patients will be attending together. After the individual BHC visit and each class, patients had behavioral "homework" to complete.
  Interventions: Behavioral: Focused Acceptance & Commitment Therapy (FACT)
- Enhanced Treatment as Usual (ETAU) (Active Comparator): Patients randomized to the Enhanced-Treatment As Usual (ETAU) group received "enhancement" of usual primary care via 1-page (2-sided) educational handouts on four topic areas: Sleep, Pacing, Relaxation and Goal Setting. All topics have an evidence base in standard Cognitive Behavioral Therapy treatment of pain. One handout per assessment visit was given to each patient. Patients will continue to see their primary care clinicians and have access to all routine clinical services throughout the study.
  Interventions: Behavioral: Enhanced Treatment as Usual (ETAU)

INTERVENTIONS:
Behavioral: Focused Acceptance & Commitment Therapy (FACT) — FACT is a brief form of Acceptance and Commitment Therapy and in this study, FACT focused on increasing patient functioning through connection with valued activities and increased acceptance.
  Arms: Focused Acceptance and Commitment Therapy (FACT)
Behavioral: Enhanced Treatment as Usual (ETAU) — This active control intervention included 4 handouts focused on pain management based on cognitive behavioral science.
  Arms: Enhanced Treatment as Usual (ETAU)

SUMMARY:
This mixed-methods pilot randomized controlled trial sought to: 1) evaluate implementation of a brief Acceptance and Commitment Therapy treatment for chronic pain delivered by an integrated behavioral health consultant in primary care; and to 2) explore treatment outcomes and their associated mechanisms of change.

DETAILED DESCRIPTION:
Background: Most patients with chronic pain obtain their treatment in primary care settings, where evidence-based behavioral interventions are not typically provided, despite robust evidence for treatments like Acceptance and Commitment Therapy.

Objective: This mixed-methods pilot randomized controlled trial sought to: 1) evaluate implementation of a brief Acceptance and Commitment Therapy treatment for chronic pain delivered by an integrated behavioral health consultant in primary care; and to 2) explore treatment outcomes and their associated mechanisms of change.

Design: Mixed-methods pilot randomized controlled trial. Active participants completed one 30-minute individual Focused Acceptance and Commitment Therapy (FACT) visit followed by 3 weekly 60-minute group visits and a booster visit 2 months later. An enhanced treatment as usual (ETAU) control group received 4 handouts about pain management based on cognitive behavioral science. Follow-up research visits occurred during and after treatment, at 12 weeks (booster visit), and at 6 months. Semi-structured interviews were conducted after the last research visit.

Setting: A small integrated primary care clinic in southwestern U.S. affiliated with an academic medical center

ELIGIBILITY:
Inclusion Criteria:

* age 18 and older
* at least one non-cancer pain condition persisting for 12 weeks or more
* a current primary care clinician at the study clinic
* ongoing treatment for a non-cancer chronic pain condition

Exclusion Criteria:

* social anxiety or unwillingness to participate in a class setting
* presence of symptoms of psychosis and/or delirium
* a medical condition or life circumstance that would contraindicate or prevent participating (e.g. upcoming surgery)
* inability to comprehend the informed consent process or study instructions.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2017-10-09 (Actual); Primary Completion 2018-12-10 (Actual); Study Completion 2019-04-22 (Actual)

PRIMARY OUTCOMES:
Self-reported physical disability | Booster (12 weeks from baseline)
  The Oswestry Disability Index (ODI) is a 10-item self-report scale that assesses perceived disability and functional impairment across a range of daily activities, with higher scores indicating greater perceived disability. Although originally developed as a measure of back pain, we used an established modified version that asked about "pain" rather than "back pain." The ODI uses a 6-point Likert scale for each item, which is summed to create a total score (maximum 50) that is then divided by highest possible score based on items skipped, and doubled to provide a percentage of patient perceived disability. The ODI and has been validated across a wide range of populations as a reliable and useful indicator of overall disability. Scores range from 0-100.
Self-reported physical disability | 6-month follow-up
  The Oswestry Disability Index (ODI) is a 10-item self-report scale that assesses perceived disability and functional impairment across a range of daily activities, with higher scores indicating greater perceived disability. Although originally developed as a measure of back pain, we used an established modified version that asked about "pain" rather than "back pain." The ODI uses a 6-point Likert scale for each item, which is summed to create a total score (maximum 50) that is then divided by highest possible score based on items skipped, and doubled to provide a percentage of patient perceived disability. The ODI and has been validated across a wide range of populations as a reliable and useful indicator of overall disability. Scores range from 0 - 100.
Feasibility of intervention and study (attrition and satisfaction ratings) | 6-month follow-up
  Feasibility was evaluated using a priori established benchmarks: (a) < 25% participant attrition; (b) at least 80% of participants rating the FACT program as satisfactory as measured by response of at least 5 on a 7-point Likert-scale (1= Not Satisfied at All, 7 = Very Satisfied). The satisfaction question was asked in the context of an "exit interview": all participants who completed the 6-month follow-up assessment were contacted by the PI to provide feedback on their experiences in the study.
Acceptability of the FACT intervention | 6-month follow-up
  Acceptability of the FACT intervention from the participants' perspective was measured via 3 Likert-scale questions gathered during the semi-structured interview focused on: perceived benefit, ease of learning about pain management, and whether the participant would recommend the FACT treatment to a friend or family member

SECONDARY OUTCOMES:
Chronic Pain Acceptance | Booster (12 weeks from baseline)
  The 20-item Chronic Pain Acceptance Questionnaire (CPAQ) assesses the degree to which activities are done in the presence of chronic pain and pain-related experiences (Activities Engagement), and the degree of effort put in to controlling pain (Willingness). Each of the 20 items uses a 6-point numerical rating scale. The CPAQ has acceptable psychometrics in many studies and each item uses a 6-point numerical rating scale. There are no established cut-points, although higher scores on the CPAQ indicate greater acceptance of chronic pain. Scores range from 0 - 120.
Chronic Pain Acceptance | 6-month follow-up
  The 20-item Chronic Pain Acceptance Questionnaire (CPAQ) assesses the degree to which activities are done in the presence of chronic pain and pain-related experiences (Activities Engagement), and the degree of effort put in to controlling pain (Willingness). Each of the 20 items uses a 6-point numerical rating scale. The CPAQ has acceptable psychometrics in many studies and each item uses a 6-point numerical rating scale. There are no established cut-points, although higher scores on the CPAQ indicate greater acceptance of chronic pain. Scores range from 0 - 120.
Engagement in Valued Activities | Booster (12 weeks from baseline)
  The Chronic Pain Values Inventory (CPVI) identifies which values are important to a person with chronic pain, and assesses the degree of success they are having in following their values. The valued domains are family, intimate relations, friends, work, health, and growth or learning. The 12-item CPVI uses 6-point Likert scale questions to measure the discrepancy between ratings of importance of valued life areas and success in engaging in those life areas; lower scores reflect greater alignment (i.e., less discrepancy) between values and actions in one's life. Scores range from 0-6.
Engagement in Valued Activities | 6-month follow-up
  The Chronic Pain Values Inventory (CPVI) identifies which values are important to a person with chronic pain, and assesses the degree of success they are having in following their values. The valued domains are family, intimate relations, friends, work, health, and growth or learning. The 12-item CPVI uses 6-point Likert scale questions to measure the discrepancy between ratings of importance of valued life areas and success in engaging in those life areas; lower scores reflect greater alignment (i.e., less discrepancy) between values and actions in one's life. Scores range from 0-6.

CONTACTS AND LOCATIONS:
Overall Officials: Kathryn Kanzler, Principal Investigator — University of Texas Health San Antonio
Locations (1):
- Medical Drive Primary Care, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
The data that support the findings of this study are available from the corresponding author, [author initials], upon reasonable request
Supporting Information: Study Protocol, SAP, ICF, CSR

REFERENCES:
- [Derived] Kanzler KE, Robinson PJ, McGeary DD, Mintz J, Kilpela LS, Finley EP, McGeary C, Lopez EJ, Velligan D, Munante M, Tsevat J, Houston B, Mathias CW, Potter JS, Pugh J. Addressing chronic pain with Focused Acceptance and Commitment Therapy in integrated primary care: findings from a mixed methods pilot randomized controlled trial. BMC Prim Care. 2022 Apr 14;23(1):77. doi: 10.1186/s12875-022-01690-2. PMID 35421949